CLINICAL TRIAL: NCT01849484
Title: Effect of Hippocampal Sparing on Neurocognitive Functions and Quality of Live in Patients Irradiated in the Neurocranial Area
Brief Title: Enhancement of Neurocognitive Functions by Hippocampal Sparing Radiotherapy
Acronym: HIPPO-SPARE 01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIPSPA2013
Record Dates: First submitted 2013-05-03; First posted 2013-05-08 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Radiation of Neurocranial Region
Keywords: meningioma; skull base meningioma; pituitary adenoma; brain metastases; small cell lung carcinoma
MeSH Terms: conditions — Meningioma; Pituitary Neoplasms; Brain Neoplasms; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hippocampal sparing radiotherapy (Experimental): Radiation according to indication with hippocampal sparing
  Interventions: Radiation: Radiation according to indication with hippocampal sparing
- Control (Active Comparator): Radiation according to indication without hippocampal sparing
  Interventions: Radiation: Radiation according to indication without hippocampal protection

INTERVENTIONS:
Radiation: Radiation according to indication with hippocampal sparing — Performed with hippocampal sparing Meningioma-total dose up to 50.4 Gy (+ additional boost up to 59.4 Gy) Hypophyseal adenoma - total dose up to 50.4 Gy (+additional boost up to 54 Gy) SCLC (prophylactic cranial irradiation) - total dose up to 36.0 Gy
  Arms: hippocampal sparing radiotherapy
Radiation: Radiation according to indication without hippocampal protection — Performed with hippocampal sparing Meningioma-total dose up to 50.4 Gy (+ additional boost up to 59.4 Gy) Hypophyseal adenoma - total dose up to 50.4 Gy (+additional boost up to 54 Gy) SCLC (prophylactic cranial irradiation) - total dose up to 36.0 Gy
  Arms: Control

SUMMARY:
This randomized trial examines possible enhancements in live quality and neurocognitive functions in patients after radiotherapy of the neurocranial area with hippocampal sparing. Although the hippocampus has a crucial role in regard to neurocognition and memory, hippocampal region has been relatively disregarded in radiotherapy of neurocranium so far. Brain metastases in the hippocampal region are very rare and an infiltration of the hippocampus by meningioma or by pituitary adenoma just occurs when volume of the tumor is very high. This study aims to reduce the radiation dose in the hippocampal region to improve the quality of live and neurocognitive functions in patients without degrading prognosis or increasing probability of brain metastases in hippocampal region.

Primary endpoint of the trial is quality of live and neurocognitive functions in patients after radiation of neurocranial region with hippocampal sparing compared with conventional radiotherapy of the neurocranial region without hippocampal sparing. Secondary endpoints are cerebral recurrence rate in hippocampal region and overall survival. It is planned to include a total number of 150 patients.

ELIGIBILITY:
Inclusion Criteria:

* minimum age 18
* diseases indicating a radiotherapy of neurocranial area (histologically or image-guided confirmed (skull base)meningioma,pituitary adenoma,brain metastases, SCLC)
* indication for a local radiotherapy in neurocranial area or for a radiation of whole neurocranium
* Karnofsky-State ≥ 50%
* patient has understand content of study protocol
* Signed study-specific consent form prior to therapy

Exclusion Criteria

* pregnant or nursing women
* Fertile patients who refuse effective contraception during study treatment
* persistent drug and/or alcohol abuse
* prior radiotherapy of neurocranial region
* patients not able or willing to behave according to study protocol
* in the case of malignancy: more than 3 brain metastases
* in the case of malignancy: brain metastases in hippocampal region or in the hippocampus avoidance zone
* GTV in hippocampal region or in the hippocampus avoidance zone
* patients in care
* patients who are not able to speak German
* conditions that preclude the application of MRT (e.g. magnetic implants, cardiac pacemaker)
* on-treatment participation on other trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-03; Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
quality of live and neurocognitive functions | Participants will be followed for the duration of therapy and for 5 years after the last study treatment

SECONDARY OUTCOMES:
cerebral recurrence rate in hippocampal region | Participants will be followed for the duration of therapy and for 5 years after the last study treatment
overall survival | Participants will be followed for the duration of therapy and for 5 years after the last study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Fietkau, MD, Principal Investigator — Strahlenklinik, Universitätsklinikum Erlangen
Locations (1):
- Universitätsklinikum Erlangen, Erlangen, Germany